CLINICAL TRIAL: NCT05647655
Title: Value of Transthoracic Ultrasonography (TTU) for Etiological Diagnosis of Acute Dyspnea: Cross Sectional Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Alaa Eldin Abd El Moniem, Principal Investigator, Assiut University
Other Study IDs: US in Acute dyspnea
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2022-12

CONDITIONS: Dyspnea
MeSH Terms: conditions — Dyspnea | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasonography — Bedside thoracic ultrasound for patients complaining of acute dyspnea.

SUMMARY:
Evaluating the capability and efficiency of transthoracic ultrasound in attempting to identify the etiology of acute dyspnea.

DETAILED DESCRIPTION:
Acute dyspnea is a frequent challenge for physicians due to having multiple etiologies, leading to difficulty in establishing an accurate diagnosis.

The presence of this symptom is already a predictor of increased mortality and a lot of investigations are required to differentiate between etiologies. Hence, prompt diagnosis is needed to streamline these patients' appropriate management and disposition from the ED.

Transthoracic ultrasound has traditionally been used for the detection of pleural effusion and evaluation of the chest wall, but the indications have been expanded.

The gold standard imaging technique for the majority of pulmonary disorders is high-resolution computed tomography (HRCT), but it has negatives which are:

* hazard of ionizing radiation
* high cost
* being nonportable

ELIGIBILITY:
Inclusion Criteria:

* Clinical history of acute dyspnea

Exclusion Criteria:

* Subcutaneous emphysema.
* Patients with more than 24 h interval between HRCT and TTU.
* Patients with poor-quality of TTU image.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years with acute dyspnea will be included
Sampling Method: Probability Sample
Enrollment: 143 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Differentiate between different etiologies of acute dyspnea | Baseline
  Analysis of ultrasound findings to differentiate between etiologies of acute dyspnea.

SECONDARY OUTCOMES:
Detect value of transthoracic ultrasound (TTU) in comparison to CT chest. | Baseline
  Comparison between accuracy of TTU and CT

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Elsayed, MBBCH, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Egypt

REFERENCES:
- [Background] Gargani L, Fontana M, Sicari R, Picano E. [Differential diagnosis of dyspnea: the incremental value of lung ultrasound]. Recenti Prog Med. 2010 Feb;101(2):78-82. Italian. PMID 20433006
- [Background] Baid H, Vempalli N, Kumar S, Arora P, Walia R, Chauhan U, Shukla K, Verma A, Chawang H, Agarwal D. Point of care ultrasound as initial diagnostic tool in acute dyspnea patients in the emergency department of a tertiary care center: diagnostic accuracy study. Int J Emerg Med. 2022 Jun 13;15(1):27. doi: 10.1186/s12245-022-00430-8. PMID 35698060
- [Background] Vitturi N, Soattin M, Allemand E, Simoni F, Realdi G. Thoracic ultrasonography: A new method for the work-up of patients with dyspnea(). J Ultrasound. 2011 Sep;14(3):147-51. doi: 10.1016/j.jus.2011.06.009. Epub 2011 Jun 30. PMID 23396858
- [Background] Li H, Li YD, Zhu WW, Sun LL, Ye XG, Kong LY, Cai QZ, Jiang W, Wang L, Lu XZ. High-Resolution Transthoracic Ultrasonography for Assessment of Pleural Lines in Patients With Dyspnea With CT Comparison: An Observational Study. J Ultrasound Med. 2017 Apr;36(4):707-716. doi: 10.7863/ultra.16.04030. Epub 2017 Jan 27. PMID 28127786
- [Background] Lancellotti P, Price S, Edvardsen T, Cosyns B, Neskovic AN, Dulgheru R, Flachskampf FA, Hassager C, Pasquet A, Gargani L, Galderisi M, Cardim N, Haugaa KH, Ancion A, Zamorano JL, Donal E, Bueno H, Habib G. The use of echocardiography in acute cardiovascular care: recommendations of the European Association of Cardiovascular Imaging and the Acute Cardiovascular Care Association. Eur Heart J Cardiovasc Imaging. 2015 Feb;16(2):119-46. doi: 10.1093/ehjci/jeu210. Epub 2014 Nov 6. PMID 25378470